CLINICAL TRIAL: NCT06777784
Title: An In-Clinic Confinement Study to Assess Elements of Abuse Liability for Six Modern Nicotine Oral Products
Brief Title: Modern Nicotine Oral Product Abuse Liability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RAI Services Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CSD241801
Record Dates: First submitted 2025-01-10; First posted 2025-01-16 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Smoking; Tobacco Use
MeSH Terms: conditions — Smoking; Tobacco Use | interventions — HTR3D protein, human

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Product usage order ANBGCFDE (Experimental): Subjects will use each of the 8 products during an evaluation period, followed by a 4 hour Test Session
  Interventions: Other: Product A; Other: Product B; Other: Product C; Other: Product D; Other: Product E; Other: Product F; Other: Product G; Other: Product N
- Product usage order BACNDGEF (Experimental): Subjects will use each of the 8 products during an evaluation period, followed by a 4 hour Test Session
  Interventions: Other: Product A; Other: Product B; Other: Product C; Other: Product D; Other: Product E; Other: Product F; Other: Product G; Other: Product N
- Product usage order CBDAENFG (Experimental): Subjects will use each of the 8 products during an evaluation period, followed by a 4 hour Test Session
  Interventions: Other: Product A; Other: Product B; Other: Product C; Other: Product D; Other: Product E; Other: Product F; Other: Product G; Other: Product N
- Product usage order DCEBFAGN (Experimental): Subjects will use each of the 8 products during an evaluation period, followed by a 4 hour Test Session
  Interventions: Other: Product A; Other: Product B; Other: Product C; Other: Product D; Other: Product E; Other: Product F; Other: Product G; Other: Product N
- Product usage order EDFCGBNA (Experimental): Subjects will use each of the 8 products during an evaluation period, followed by a 4 hour Test Session
  Interventions: Other: Product A; Other: Product B; Other: Product C; Other: Product D; Other: Product E; Other: Product F; Other: Product G; Other: Product N
- Product usage order FEGDNCAB (Experimental): Subjects will use each of the 8 products during an evaluation period, followed by a 4 hour Test Session
  Interventions: Other: Product A; Other: Product B; Other: Product C; Other: Product D; Other: Product E; Other: Product F; Other: Product G; Other: Product N
- Product usage order GFNEADBC (Experimental): Subjects will use each of the 8 products during an evaluation period, followed by a 4 hour Test Session
  Interventions: Other: Product A; Other: Product B; Other: Product C; Other: Product D; Other: Product E; Other: Product F; Other: Product G; Other: Product N
- Product usage order NGAFBECD (Experimental): Subjects will use each of the 8 products during an evaluation period, followed by a 4 hour Test Session
  Interventions: Other: Product A; Other: Product B; Other: Product C; Other: Product D; Other: Product E; Other: Product F; Other: Product G; Other: Product N

INTERVENTIONS:
Other: Product A — Usual Brand (UB) filtered, menthol or non-menthol combustible cigarette
Other: Product B — Modern Nicotine Oral Product Cool Mint 6 mg Nicotine
Other: Product C — Modern Nicotine Oral Product Cool Mint 12 mg Nicotine
Other: Product D — Modern Nicotine Oral Product Cool Mint 15 mg Nicotine
Other: Product E — Modern Nicotine Oral Product Smooth 6 mg Nicotine
Other: Product F — Modern Nicotine Oral Product Wintergreen 6 mg Nicotine
Other: Product G — Modern Nicotine Oral Product Dragon Fruit 6 mg Nicotine
Other: Product N — Nicorette® White Ice Mint 4 mg nicotine gum

SUMMARY:
This is a two-site, open-label, randomized, 8-way cross-over study designed to evaluate elements of abuse liability (AL) including subjective effects and physiological measures (pharmacodynamics [PD]) and plasma nicotine uptake (pharmacokinetics [PK]) during and following ad libitum use of the study investigational products (IPs) by generally healthy smokers.

DETAILED DESCRIPTION:
Cigarette smokers naïve to smokeless tobacco products (ST) and smokers also using ST will be recruited into this AL study to evaluate elements of AL of six modern oral nicotine products compared to combustible cigarettes (CC) and nicotine polacrilex gum. An attempt will be made for at least one-third of the study population to include smokers using ST.

Potential subjects will complete a pre-screening telephone interview. They will complete a Screening Visit to assess their eligibility within 45 days prior to check-in and enrollment.

Starting on check in day (Day -1), subjects will check-in at the clinical site to complete procedures to confirm eligibility. Eligible subjects will be enrolled, randomized and confined for 10 days (9 nights). Prior to the first product acclimation period, subjects will conduct a product familiarization of three of the modern oral nicotine products. Subjects will be randomized to one of eight product use sequences (using a Williams Design) in which they will evaluate one IP in each of eight separate Test Sessions, such that each subject will evaluate eight IPs, including six modern oral nicotine products, and both a high-AL comparator (subject's usual brand [UB] cigarette) and a low-AL comparator (a commercially available nicotine replacement therapy [NRT] nicotine gum).

On Day 2 and continuing through Day 9, subjects will participate in Test Sessions that will last approximately 4 hours. Each Test Session will include collection of both types of PD measures (subjective and physiological) and PK measures prior to, during, and following IP use.

On the half day prior to each respective Test Session, a Product Acclimation Period will allow subjects ad libitum use of the subsequent IP (at least two trial uses) as per randomized sequence for product acclimation prior to use in the next day's Test Session. Subjects can also use their UB cigarettes ad libitum, until the 12-hour tobacco and nicotine abstinence period begins prior to each Test Session, as long as the minimum use requirement for randomized IP is met.

ELIGIBILITY:
Inclusion Criteria:

1. Able to read, understand, and willing to sign an informed consent form (ICF) and complete questionnaires written in English.
2. Generally healthy males or females, 21 to 60 years of age, inclusive, at the time of consent.
3. Smokes combustible, filtered, non-menthol or menthol cigarettes, 83 mm to 100 mm in length as primary source of tobacco.
4. Smokes an average of at least 10 cigarettes per day (CPD) and inhales the smoke, for at least 6 months prior to Screening. Brief periods of abstinence due to illness, quit attempt (prior to 30 days of Screening), or clinical study participation (prior to 30 days of Screening) will be allowed at the discretion of the an investigator.
5. Smokers who also use ST products (e.g., moist snuff, snus, modern oral), and have used ST within 30 days prior to screening, will be enrolled.
6. Agrees to smoke the same UB cigarette throughout the study period. The UB cigarette is defined as the reported cigarette brand and style currently smoked most frequently by the subject.
7. Expired breath carbon monoxide (ECO) level is ≥ 10 ppm and ≤ 100 ppm at Screening and at check-in (Day -1).
8. Positive urine cotinine test (e.g., >200 ng/mL) via dipstick at Screening.
9. Response at Screening to the Fagerström Test for Nicotine Dependence (FTND) Question 1 ("How soon after you wake up do you smoke your first cigarette?") is either "Within 5 minutes" or "6-30 minutes" (Heatherton et al., 1991).
10. Willing to use the UB cigarette, Velo PLUS IPs, and Nicorette® nicotine gum during the study period.
11. Willing to abstain from tobacco and nicotine use for at least 12 hours prior to the start of each of eight Test Sessions.
12. Females must be willing to use a form of contraception acceptable to an investigator from the time of signing the ICF until End-of-Study. Examples of acceptable means of birth control are, but not limited to: a) Surgical sterilization (hysterectomy, bilateral tubal ligation/occlusion, bilateral oophorectomy, bilateral salpingectomy); b) physical barrier method (e.g., condom, diaphragm/sponge/cervical cap) with spermicide; c) non-hormone releasing intrauterine devices (IUD) or hormone-releasing IUDs (e.g., Mirena or Kyleena); d) vasectomized partner; or e) post-menopausal and not on hormone replacement therapy.
13. Agrees to an in-clinic confinement of ten days (nine nights).

Exclusion Criteria:

1. Allergic to or cannot tolerate mint or wintergreen flavoring agents.
2. Individuals or their family members that have ongoing litigation with tobacco company(ies)
3. Have used electronic nicotine delivery system (e.g., Vuse Alto, JUUL) or tobacco heating device (e.g., iQOS) within the last 30 days prior to screening.
4. Presence of clinically significant uncontrolled cardiovascular, pulmonary, renal, hepatic, endocrine, gastrointestinal, psychiatric, hematological, neurological disease, or any other concurrent disease or medical condition that, in the opinion of an investigator, makes the study subject unsuitable to participate in this clinical study.
5. History, presence of, or clinical laboratory test results indicating diabetes.
6. Scheduled treatment for asthma currently or within the past consecutive 12 months prior to the Screening Visit. As-needed treatment, such as inhalers, may be included at an investigator discretion.
7. History or presence of bleeding or clotting disorders.
8. Any history of cancer, except for primary cancers of skin such as localized basal cell/squamous cell carcinoma that has been surgically and/or cryogenically removed.
9. Systolic blood pressure of > 160 mmHg or a diastolic blood pressure of > 95 mmHg, measured after being seated for five minutes at Screening or at check-in Day -1.
10. Weight of ≤ 110 pounds at screening or at check-in.
11. Hemoglobin level is < 12.5 g/dL for females or < 13.0 g/dL for males at Screening.
12. Females who have a positive pregnancy test, are pregnant, breastfeeding, or intend to become pregnant during the course of the study.
13. Has positive urine drug screen (UDS) or alcohol test (urine or breath) at Screening or at Check-in to the Assessment Phase (Day -1), with the exception of positive results for tetrahydrocannabinol (THC). If positive for THC at check-in (Day -1), a cannabis intoxication evaluation will be performed, and inclusion will be at the discretion of an investigator.
14. Positive test for human immunodeficiency virus (HIV), hepatitis B surface antigen (HbsAg), or hepatitis C virus (HCV).
15. Use of any medication or substance that aids in smoking cessation, including but not limited to any NRT (e.g., nicotine gum, lozenge, patch), varenicline (Chantix®), bupropion (Wellbutrin®, Zyban®), or lobelia extract within (≤) 30 days prior to signing the informed consent.
16. Postpones a decision to quit using tobacco- or nicotine-containing products in order to participate in this study or self-reports a previous quit attempt within (≤) 30 days prior to signing the informed consent.
17. Any use of daily aspirin (≥ 325 mg) or any use of other anticoagulants.
18. Individuals ≥ 35 years of age currently using systemic, testosterone, estrogen-containing contraception or hormone replacement therapy.
19. Whole blood donation or lost blood or blood products in excess of 500 mL within 8 weeks (≤ 56 days) prior to signing the informed consent and between Screening and check-in Day -1.
20. Plasma donation within (≤) 7 days prior to signing the informed consent and between Screening and check-in Day -1.
21. Employed by a tobacco or nicotine company, the study site, or handles raw, unpackaged tobacco- or nicotine-containing products as part of their job.
22. Has used an investigational drug, device, biologic, or tobacco/nicotine product in a previous clinical study within 30 days or 5 times the half-life of the product (whichever is longer) prior to Screening.
23. Drinks more than 21 servings of alcoholic beverages per week.
24. Determined by an investigator to be inappropriate for this study.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2025-02-03 (Actual); Primary Completion 2025-03-05 (Actual); Study Completion 2025-03-05 (Actual)

PRIMARY OUTCOMES:
AUECPL 5-240 | 5 minutes to 240 minutes
  area under the effect curve (AUEC) for PL (VAS score-versus-time)
Emax PL | 240 minutes
  maximum effect (maximum PL VAS score after the start of IP use)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Keyser, PhD, Study Director — Reynolds American
Locations (2):
- United States (2):
  - AMR Lexington, Lexington, Kentucky
  - AMR Knoxville, Knoxville, Tennessee

IPD SHARING:
Plan to Share IPD: No